CLINICAL TRIAL: NCT07371156
Title: Patient-centred Modular Cognitive Behavioural Therapy Versus Prolonged Exposure Therapy for Complex Post-traumatic Stress Disorder: a Randomised Trial
Brief Title: PACE Versus PE for CPTSD (PACE Trial)
Acronym: PACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sofie Folke (Other Government)
Collaborators: Danish Veterans Centre (Other Government); Aarhus University Hospital (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor-Investigator, Sofie Folke, PhD, Psychologist, Senior Researcher, Danish Veterans Centre
Organization: Danish Veterans Centre (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PACE trial; H-25066014 (Other: The Regional Ethics Committees, Capital Region of Denmark)
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Complex Posttraumatic Stress Disorder

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, multi-centre, parallel group, randomised clinical superiority trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors, data managers, statisticians, and conclusion drawers will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACE (Experimental): Patient-centred Modular Cognitive Behavioural Therapy
  Interventions: Other: PACE
- PE (Active Comparator): Prolonged Exposure therapy
  Interventions: Other: PE

INTERVENTIONS:
Other: PACE — 26 hours PACE (delivered as 26 1-hour sessions of weekly individual psychotherapy).
  Arms: PACE
Other: PE — 25.5 hours PE therapy (17 sessions of weekly individual psychotherapy delivered for 90-minutes).
  Arms: PE

SUMMARY:
The objective of this pragmatic trial is to evaluate the beneficial and harmful effects of Patient-centred Modular Cognitive Behavioural Therapy (PACE) compared with the standard post-traumatic stress disorder (PTSD) treatment, Prolonged Exposure (PE), for adults with an ICD-11 diagnosis of Complex post-traumatic stress disorder (CPTSD).

DETAILED DESCRIPTION:
This trial is designed as an investigator-initiated, multi-centre, parallel group, randomised clinical superiority trial of PACE versus standard PTSD treatment, PE, for ICD-11 CPTSD. The total sample size will be 228 participants. The trial will take place at the Danish Veteran Centre and two clinics in the Mental Health Services in Denmark. The participants will be adult military veterans and psychiatric outpatients with ICD-11 CPTSD. After giving their consent, participants will be randomly assigned (1:1) to receive either PACE or PE.

The experimental intervention will be 26 hours PACE (delivered as 26 1-hour sessions of weekly individual psychotherapy). The control intervention will be 25.5 hours PE therapy (17 sessions of weekly individual psychotherapy delivered for 90-minutes).

Outcome assessors, data managers, statisticians, and conclusion drawers will be blinded to group allocation. The primary outcome will be clinician-rated ICD-11 CPTSD symptom severity assessed with the International Trauma Interview (ITI) at 9 months after randomisation. Secondary outcomes include serious adverse events, suicide attempts, symptoms of depression, stress, and anxiety, alcohol use problems, mental well-being, and functional impairment assessed at 9 months after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years.
* Referred to PTSD treatment (which requires absence of severe psychiatric comorbidity dominating the clinical presentation, hindering trauma-focused psychotherapy, assessed by the referring clinician at point of referral (e.g. major depressive disorder, ADHD, autism spectrum disorders, personality disorders, psychotic disorders, alcohol- or substance use, and aggressive behaviours)).
* Diagnosis of CPTSD according to ICD-11, assessed by the interviewing investigator using the ITI interview.
* Written informed consent.

Exclusion Criteria:

* Current self-harm or severe suicidality defined as at least one self-harm episode or one suicide-attempt the last three months, as assessed by the interviewing investigator.
* Any other condition that markedly compromises the participant's ability to adhere to the treatment programme or follow-up, such IQ < 70 based on clinical judgement.
* Currently involved in legal proceedings concerning work accident compensation related to PTSD, or trial regarding child custody.
* Does not understand Danish or needs an interpreter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
ITI | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  CPTSD symptom severity assessed with the International Trauma Interview (ITI), (scale ranging from 0-48, higher scores indicate higher severity)

SECONDARY OUTCOMES:
SAE | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Proportion of participants with at least one serious adverse event (SAE) during the intervention period, assessed via patient medical records by a blinded outcome adjudication committee. SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalisation or prolonging of existing hospitalisation, and resulted in persistent or significant disability or jeopardised the participant.
Suicides and suicide attempts | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Proportion of participants with a suicide- or a suicide attempt during the intervention period, assessed via patient medical records by a blinded outcome adjudication committee.
DASS-21, depression | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Symptoms of depression, assessed using the depression subscale from the Depression Anxiety Stress Scales-21 items (DASS-21), (scale ranging from 0-42, higher scores indicate higher severity of depression symptoms).
DASS-21, anxiety | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Symptoms of anxiety, assessed using the anxiety subscale from the Depression Anxiety Stress Scales-21 items (DASS-21), (scale ranging from 0-42, higher scores indicate higher severity of anxiety symptoms).
AUDIT | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Alcohol use problems, assessed using the Alcohol Use Disorders Identification Test (AUDIT), (scale from 0-40, higher scores indicate greater risk).
WHO-5 | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Mental well-being, assessed using the World Health Organization-Five Well-Being Index (WHO-5), (percentage score from 0-100, higher scores indicate better well-being).
SDS | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Level of functioning, assessed using the Sheehan Disability Scale (SDS), (scale ranging from 0 (unimpaired) to 30 (highly impaired)).

OTHER OUTCOMES:
ITQ | 3, 6, and 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Symptoms of ICD-11 complex PTSD, assessed with the International Trauma Questionnaire (ITQ), (a total symptom severity score will be calculated by summing PTDS items (P1-P6) and Disturbances in Self-Organization (items C1-C6) symptoms, yielding a score ranging from 0-48, with higher scores indicating greater CPTSD symptom severity)
TIQ | 3, 6, and 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Trauma-related identity, assessed with the Trauma Identity Questionnaire, (scale ranging from 0 to 105 with higher scores representing presence of negative identity characteristics associated with traumatic experiences).
ETMQ | 3, 6, and 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Sensory and cognitive-emotional qualities of traumatic memories, assessed with the Experiences of Traumatic Memories Questionnaire (ETMQ), (scores range from 0-32 with higher scores reflecting more intense sensation-based trauma memories).
CSS | 3, 6, and 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Level of perceived social support, assessed with the Crisis Support Scale (CSS), (scale ranging from 6-42, higher scores indicate greater perceived social support).
EQ-5D-5L | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Health-related quality of life, assessed using the European Quality of Life - 5 Dimensions, 5 Levels (EQ-5D-5L). Index score (score between -1 and 1, higher scores indicate better health).
DSS | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Dissociative symptoms, assessed using the Dissociative Symptoms Scale (DSS), Scale ranging from 0 to 80, higher scores indicate greater dissociative symptom severity).
MIOS | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Moral injury-related distress, assessed using the Moral Injury Outcome Scale (MIOS), (scale ranging from 0 to 56, higher scores indicate greater moral injury-related distress).
ISI | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Insomnia severity, assessed using the Insomnia Severity Index (ISI), (scale ranging from 0 (no problem) to 28 (severe insomnia)).
DASS-21, stress | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Symptoms of stress, assessed using the stress subscale from the Depression Anxiety Stress Scales-21 items (DASS-21), (scale ranging from 0-42, higher scores indicate higher severity of stress symptoms).
DUDIT | End of intervention, 9 months after randomisation (and assessed as an exploratory outcome at 18 months after randomisation)
  Drug use problems, assessed using the Drug Use Disorders Identification Test (DUDIT), (scale from 0-44, higher scores indicate greater risk of drug-related disorders).

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Folke, Principal Investigator — Military Psychology Department, Danish Veterans Centre, part of Defence Command Denmark
Locations (10):
- Denmark (10):
  - The Outpatient Clinic for PTSD, Department of Affective Disorders, Aarhus University Hospital Psychiatry, Aarhus
  - The Outpatient Clinic for PTSD at Ballerup, Mental Health Centre Ballerup, Capital Region of Denmark, Ballerup Municipality
  - Danish Veterans Centre - Høvelte: Livgardens Kaserne, Høveltevej 117, Birkerød
  - Danish Veterans Centre - Svanemøllen: Svanemøllens Kaserne, Ryvangs Allé 1-3, Copenhagen
  - Danish Veterans Centre - Fredericia: Ryes Kaserne, Treldevej 110, Fredericia
  - Danish Veterans Centre - Holstebro: Jydske Dragonregiment, Dragonkasernen 1, Holstebro
  - Danish Veterans Centre - Karup: Flyvestation Karup, Herningvej 30, Karup
  - Danish Veterans Centre - Aalborg: Aalborg Kaserner, Gl. Høvej 34, Nørresundby
  - Danish Veterans Centre - Ringsted: Ringsted Kaserne, Garnisonen 1, Ringsted
  - Danish Veterans Centre - Slagelse: Antvorskov Kaserne, Charlottedal Allé 4, Slagelse

IPD SHARING:
Plan to Share IPD: Yes
After the results have been published, we aim to make a depersonalised dataset publicly available on e.g. ClinicalTrials.gov and/or the European Union (EU) Zenodo database (https://zenodo.org/). The final choice will reflect which platform(s) that are compliant with current legislation at that time.
Supporting Information: Study Protocol, SAP
Time Frame: When the results have been published.
Access Criteria: Researchers with a protocol for their planned study.